CLINICAL TRIAL: NCT05160025
Title: Enhancing Exercise Intensity, Motivation and Enjoyment for Persons With PD (VCycle-Competition)
Brief Title: Immersive Virtual Reality Bicycling for Persons With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Judith E Deutsch, PT, PhD, Professor, Department of Rehabilitation & Movement Sciences, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro2021001412; 1F30AG072807-01 (NIH); 1R15AG063348-01 (NIH)
Record Dates: First submitted 2021-10-26; First posted 2021-12-16 (Actual); Results first posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Parkinson Disease
Keywords: parkinson disease; parkinsonian disorders; Basal ganglia disease; Brain diseases; central nervous system diseases; nervous system diseases; movement disorders; synucleinopathies; neurodegenerative diseases
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders; Basal Ganglia Diseases; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Movement Disorders; Synucleinopathies; Neurodegenerative Diseases

STUDY DESIGN:
Intervention Model Description: Repeated measures design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Bicycling (Other): This is a single arm study in which all participants will execute the same three bicycling tasks over one session. Exercise intensity and enjoyment are measured while participants bicycle in a virtual reality environment (wearing virtual reality goggles) in three different conditions lasting approximately 8 minutes each.
  Interventions: Other: Virtual reality bicycling

INTERVENTIONS:
Other: Virtual reality bicycling — This is a single arm study in which all participants will execute the same three bicycling tasks over one session. Exercise intensity and enjoyment are measured while participants bicycle in a virtual reality environment (wearing virtual reality goggles) in three different conditions lasting approximately 8 minutes each.

SUMMARY:
This study has three objectives about persons with Parkinson's Disease during bicycling:

1. Determine the effect of visual feedback and competition during virtual bicycling on neuromuscular and cardiovascular intensity
2. Determine the effect of visual-feedback and competition during virtual bicycling on the user experience of motivation, enjoyment & perception of exercise intensity
3. Determine if attention differs during visual feedback compared to competition virtual bicycling

DETAILED DESCRIPTION:
Participants will attend one sessions lasting about 2-3 hours. They will complete movement assessments and questionnaires about physical activity. They will then exercise exercise in three different virtual reality augmented bicycling conditions while wearing a head mounted display (goggles). Each of the three conditions will last approximately 8 minutes and will be followed by questionnaires about the participant's experience.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Parkinson's disease following the UK Brain Bank Diagnostic Criteria,
* Hoehn and Yahr stages II-III,
* 45-80 years old,
* Able to ride a stationary upright bicycle,
* Able to sign informed consent.

Exclusion Criteria:

* Have a recent history of severe heart disease, severe lung disease, uncontrolled diabetes, traumatic brain injury or neurological disorder other than Parkinson Disease,
* Are unable to follow directions or sign a consent form,
* Do not have adequate vision or hearing ability to see or hear a television,
* Have unstable medical condition or musculoskeletal disorder such as severe arthritis, recent knee surgery, hip surgery, or any other condition that the investigators determine would impair the ability to ride the bicycle,
* Have any other medical condition that prevents bicycling,
* Have moderate depression (score of 9 or more on GDS screening tool).

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith E Deutsch, Principal Investigator — Rutgers School of Health Professions
Locations (1):
- Rutgers School of Health Professions, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Immediately following completion of the proposed study the investigators will submit a de-identified data set of the protocol and links to published papers.
Supporting Information: Study Protocol
Time Frame: The investigators will make study data available immediately following completion.
Access Criteria: Open Access

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment start date: October 21, 2022
  First participant enrolled and completed study: October 27, 2022
  Recruitment end date: February 13, 2023
  Final participant enrolled and completed study: February 17, 2023
Period: Overall Study
Arm/Group | Virtual Reality Bicycling
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Of the 22 participants with PD, 21 were included in the final analyses as 1 participant was unable to complete the 3 bicycling conditions, terminating each of the 3 trials before the full 5 minutes elapsed.
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
Competitiveness (Multidimensional Competitive Orientation Inventory) [Mean (Standard Deviation); unit: units on a scale] — Competitiveness measured using 4 separate subscales of the MCOI
  units on a scale
    Self-Developmental Competitive Subscale | 4.3 (1.4)
    Hyper-Competitive Subscale | 2.0 (0.9)
    Anxious Subscale | 2.3 (1.1)
    Lack of Interest Subscale | 2.4 (1.2)
UPDRS-III Subscale [Mean (Standard Deviation); unit: units on a scale] | 40.43 (13.7)
Physical Activity Scale for the Elderly [Mean (Standard Deviation); unit: units on a scale] | 102.27 (57.03)
Geriatric Depression Scale (short form) [Mean (Standard Deviation); unit: units on a scale] | 1.29 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Neuromuscular Intensity (Bicycling Cadence, Revolutions Per Minute) - Feedback
Description: Bicycling cadence collected continuously (1 value per second, 1 Hz)
Time Frame: Session 1 - During the 8-minute feedback bout
Measure: Mean (Standard Deviation); unit: revolutions per minute (rpm)
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
revolutions per minute (rpm) | 85.44 (13.7)
Statistical Analysis 1: Comparison: Virtual Reality Bicycling; Test type: Superiority; p < 0.001, ANOVA — rmANOVA < 0.001 post hoc paired t-tests or nonparametric equivalent with correction (x3) indicated the following: self-competition > feedback (p < 0.001) other-competition > feedback (p < 0.001) self-competition = other-competition (p > 0.05)

2. Primary Outcome: Neuromuscular Intensity (Bicycling Cadence, Revolutions Per Minute) - Self-Competition
Description: Bicycling cadence collected continuously (1 value per second, 1 Hz)
Time Frame: Session 1 - During the 8-minute self-competition bout
Measure: Mean (Standard Deviation); unit: revolutions per minute (rpm)
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
revolutions per minute (rpm) | 92.97 (16.3)

3. Primary Outcome: Neuromuscular Intensity (Bicycling Cadence, Revolutions Per Minute) - Other-Competition
Description: Bicycling cadence collected continuously (1 value per second, 1 Hz)
Time Frame: Session 1 - During the 8-minute other-competition bout
Measure: Mean (Standard Deviation); unit: revolutions per minute (rpm)
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
revolutions per minute (rpm) | 93.83 (17.1)

4. Primary Outcome: Motivation (Intrinsic Motivation Inventory) - Feedback
Description: Intrinsic Motivation Inventory - enjoyment, competence, effort, and value subscales (16 questions total). Scores in each subscale are averaged, with a minimum score of 1 and a maximum score of 7. Higher scores indicate higher motivation.
Time Frame: Session 1 - Immediately after completing the 8-minute feedback bout
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
score on a scale | 6.06 [5.4 to 6.5]
Statistical Analysis 1: Comparison: Virtual Reality Bicycling; Test type: Superiority; p = 0.111, ANOVA — rmANOVA p = 0.111 post hoc paired t-tests not performed

5. Primary Outcome: Motivation (Intrinsic Motivation Inventory) - Self-Competition
Description: as for outcome 4
Time Frame: Session 1 - Immediately after completing the 8-minute self-competition bout
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
score on a scale | 6.13 (0.6)

6. Primary Outcome: Motivation (Intrinsic Motivation Inventory) - Other-Competition
Description: as for outcome 4
Time Frame: Session 1 - Immediately after completing the 8-minute other-competition bout
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
score on a scale | 6.11 (0.6)

7. Primary Outcome: Cardiovascular Intensity (Heart Rate, Beats Per Minute) - Feedback
Description: Heart rate collected continuously (1 value per second, 1 Hz)
Time Frame: Session 1 - During the 8-minute feedback bout
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 20
beats per minute (bpm) | 109.26 (9.9)
Statistical Analysis 1: Comparison: Virtual Reality Bicycling; Test type: Superiority; p < 0.001, ANOVA — rmANOVA < 0.001 post hoc paired t-tests or nonparametric equivalent corrected (x3) indicated the following: self-competition > feedback (p = 0.003) other-competition > feedback (p = 0.007) self-competition = other-competition (p > 0.05)

8. Primary Outcome: Cardiovascular Intensity (Heart Rate, Beats Per Minute) - Self-Competition
Description: Heart rate collected continuously (1 value per second, 1 Hz)
Time Frame: Session 1 - During the 8-minute self-competition bout
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 20
beats per minute (bpm) | 115.41 (12.6)

9. Primary Outcome: Cardiovascular Intensity (Heart Rate, Beats Per Minute) - Other-Competition
Description: Heart rate collected continuously (1 value per second, 1 Hz)
Time Frame: Session 1 - During the 8-minute other-competition bout
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 20
beats per minute (bpm) | 114.42 (12.4)

10. Primary Outcome: Visual Attention (Infrared Eye-tracking Data Representing Gaze Positions in a 3D Coordinate Plane to be Used in Calculating Dwell Time in Regions of Interest in the Virtual Simulation) - Feedback
Description: 3D gaze positions are measured continuously (40 values per second, 40 Hz) and valid gaze datapoints are extracted. The percentage of total valid gaze datapoints that are directed to the task are calculated as a metric of visual attention. A higher percentage reflects higher task focus, meaning that the higher percentage the higher degree of focus on the task. The reported value is measured as a percentage (%).
Time Frame: Session 1 - During the 8-minute feedback bout
Measure: Median (Inter-Quartile Range); unit: percentage of total valid gazes
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
percentage of total valid gazes | 76.70 [64.9 to 86.3]
Statistical Analysis 1: Comparison: Virtual Reality Bicycling; Test type: Superiority; p > 0.05, ANOVA — rmANOVA p > 0.05 with a partial eta squared effect size = 0.073 post hoc paired t-tests not performed

11. Primary Outcome: Visual Attention (Infrared Eye-tracking Data Representing Gaze Positions in a 3D Coordinate Plane to be Used in Calculating Dwell Time in Regions of Interest in the Virtual Simulation) - Self-Competition
Description: as for outcome 10
Time Frame: Session 1 - During the 8-minute self-competition bout
Measure: Mean (Standard Deviation); unit: percentage of total valid gazes
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
percentage of total valid gazes | 79.20 (8.8)

12. Primary Outcome: Visual Attention (Infrared Eye-tracking Data Representing Gaze Positions in a 3D Coordinate Plane to be Used in Calculating Dwell Time in Regions of Interest in the Virtual Simulation) - Other-Competition
Description: as for outcome 10
Time Frame: Session 1 - During the 8-minute other-competition bout
Measure: Mean (Standard Deviation); unit: percentage of total valid gazes
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
percentage of total valid gazes | 77.89 (9.2)

13. Secondary Outcome: Rating of Perceived Exertion - Feedback (Start)
Description: Borg scale measures a self-report of effort collected at multiple time points to compare the 3 exercise bouts. The score ranges from 6-20 with higher scores representing higher perceived exertion.
Time Frame: Session 1 - Immediately at the start (0-minute mark) of the 8-minute feedback bout
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
score on a scale | 8.43 (2.0)

14. Secondary Outcome: Rating of Perceived Exertion - Feedback (Middle)
Description: as for outcome 13
Time Frame: Session 1 - At the midpoint (4-minute mark) of the 8-minute feedback bout
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
score on a scale | 12.62 (2.3)

15. Secondary Outcome: Rating of Perceived Exertion - Feedback (End)
Description: as for outcome 13
Time Frame: Session 1 - At the endpoint (8-minute mark) of the 8-minute feedback bout
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
score on a scale | 14.0 [12.5 to 15]
Statistical Analysis 1: Comparison: Virtual Reality Bicycling; Test type: Superiority; p = 0.004, ANOVA — rmANOVA = 0.004 post hoc paired t-tests or nonparametric equivalent corrected (x3) indicated the following: self-competition > feedback (p = 0.007) other-competition > feedback (p = 0.002) self-competition = other-competition (p > 0.05)

16. Secondary Outcome: Rating of Perceived Exertion - Self-Competition (Start)
Description: as for outcome 13
Time Frame: Session 1 - Immediately at the start (0-minute mark) of the 8-minute self-competition bout
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
score on a scale | 8.67 (2.2)

17. Secondary Outcome: Rating of Perceived Exertion - Self-Competition (Middle)
Description: as for outcome 13
Time Frame: Session 1 - At the midpoint (4-minute mark) of the 8-minute self-competition bout
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
score on a scale | 13.81 (1.7)

18. Secondary Outcome: Rating of Perceived Exertion - Self-Competition (End)
Description: as for outcome 13
Time Frame: Session 1 - At the end (8-minute mark) of the 8-minute self-competition bout
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
score on a scale | 15.57 (2.0)

19. Secondary Outcome: Rating of Perceived Exertion - Other-Competition (Start)
Description: as for outcome 13
Time Frame: Session 1 - Immediately at the start (0-minute mark) of the 8-minute other-competition bout
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
score on a scale | 9.0 (2.2)

20. Secondary Outcome: Rating of Perceived Exertion - Other-Competition (Middle)
Description: as for outcome 13
Time Frame: Session 1 - At the midpoint (4-minute mark) of the 8-minute other-competition bout
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
score on a scale | 13.57 (2.5)

21. Secondary Outcome: Rating of Perceived Exertion - Other-Competition (End)
Description: as for outcome 13
Time Frame: Session 1 - At the end (8-minute mark) of the 8-minute other-competition bout
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
score on a scale | 15.0 [14 to 17.5]

22. Secondary Outcome: Competitiveness (Multidimensional Competitive Orientation Inventory)
Description: Measured once using the Multidimensional Competitive Orientation Inventory consisting of 12 items from 4 subscales (hyper competitive, self-developmental, anxious, lack of interest) For each subscale, mean scores range from 1-6 with higher scores representing higher levels of that subscale metric.
Time Frame: Measured once before exercise bouts begin (after clinical assessments) (Repeat of Baseline Outcome Measure)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
score on a scale
  Lack of Interest Subscale | 2.4 (1.2)
  Anxious Subscale | 2.3 (1.1)
  Hyper-Competitive Subscale | 2.0 (0.9)
  Self-Developmental Competitive Subscale | 4.3 (1.4)

23. Secondary Outcome: Ranking of Perceived Effort
Description: Once, after completing all 3 bicycling conditions, participants will be asked in which of the 3 bicycling conditions they felt they worked the hardest. They will rank the 3 conditions with a score from 1-3, with a 1 indicating the condition in which they felt they worked the hardest and a 3 indicating the condition in which they felt they worked the least hard.
Time Frame: Session 1 - once at the end of the session. Collected upon study completion, immediately after finishing the final bicycling condition
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
Participants
  Reported Competition against Self Condition as Most Effortful | 11
  Reported Competition against Others Condition as Most Effortful | 8
  Reported Feedback Condition as Most Effortful | 2
Statistical Analysis 1: Comparison: Virtual Reality Bicycling; Test type: Superiority; p > 0.05, Chi-squared — ranking compared to expected value for each condition and the p-value was adjusted for 3 comparisons for each condition: self-competition (p > 0.05) other-competition (p > 0.05) feedback (p > 0.05)

24. Secondary Outcome: Ranking of Enjoyment
Description: Once, after completing all 3 bicycling conditions, participants will be asked which of the 3 bicycling conditions they liked the best. They will rank the 3 conditions with a score from 1-3, with a 1 indicating the condition they liked the best and a 3 indicating the condition they liked the least.
Time Frame: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
Participants
  Liked the Competition against Self Condition the Best | 8
  Liked the Competition against Others Condition the Best | 7
  Liked the Feedback Condition the Best | 6
Statistical Analysis 1: Comparison: Virtual Reality Bicycling; Test type: Superiority; p > 0.05, Chi-squared — [p-value comment as in outcome 23, analysis 1]

25. Secondary Outcome: Audio Recordings of Exercise Experience
Description: Once, after completing all 3 bicycling conditions, participants will be asked about their exercise experience. Quantitative and qualitative analysis of recordings were not conducted. However, sample quotes representing constructs of the Intrinsic Motivation Inventory will be included in future publications.
Time Frame: as for outcome 23
Reporting Status: Not Posted

26. Other Pre Specified Outcome: UPDRS-III Subscale
Description: Description of Motor Performance Scored from 0-108 a lower score is better outcome
Time Frame: Collected once at start of the session (Repeat of Baseline Outcome Measure)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
score on a scale | 40.43 (13.7)

27. Other Pre Specified Outcome: Physical Activity Scale for the Elderly
Description: Exercise Inventory Questionnaire to measure levels of physical activity. Scores range from 0-793, and higher scores represent higher levels of physical activity over the past 7 days.
Time Frame: Collected once at start of the session (Repeat of Baseline Outcome Measure)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
score on a scale | 102.27 (57.0)

28. Other Pre Specified Outcome: Geriatric Depression Scale (Short Form)
Description: 15 item inventory to rate depression (scored from 0-15 with a lower score being better)
Time Frame: Collected once during screening (Repeat of Baseline Outcome Measure)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Reality Bicycling
Number analyzed (Participants) | 21
score on a scale | 1.29 (1.7)

ADVERSE EVENTS:
Time Frame: As this was a single session of data collection, participants were contacted the day following their data collection bicycling exercise session. Adverse event data were collected at the time of data collection and from the 1-day follow-up period.
Arm/Group | Virtual Reality Bicycling
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

LIMITATIONS AND CAVEATS:
The primary limitations are related to: setting of the baseline and target cadence, participants setting personal goals for themselves that could emulate self-competitive behavior in the competition against others condition, and operational definitions for measures of visual attention.

Other limitations: the sample of persons was recruited mostly from support groups and exercise classes in the area. Therefore, it is possible that participants were aware of the benefits of exercise.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-24): https://cdn.clinicaltrials.gov/large-docs/25/NCT05160025/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-24): https://cdn.clinicaltrials.gov/large-docs/25/NCT05160025/ICF_002.pdf